CLINICAL TRIAL: NCT01689688
Title: Healing Response to Everolimus-eluting Stent Implantation; Serial Assessment With opticaL Coherence Tomography
Acronym: HEAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kobe University (Industry)
Responsible Party: Principal Investigator, Toshiro Shinke, MD, PhD, Associate Professor, Kobe University
Other Study IDs: KobeU-001; R000008722 (Other: UMIN)
Record Dates: First submitted 2012-09-07; First posted 2012-09-21 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EES-XIENCE V: Groups who were treated with XIENCE V® everolimus eluting stent

SUMMARY:
The purpose of this study is to evaluate serial changes of neointimal coverage after everolimus-eluting stent implantation at 3-, 6- and 12-months by OCT examination.

DETAILED DESCRIPTION:
Late and very late stent thrombosis is current main issue after introduction of drug-eluting stents .Possible causes of these stent thromboses include thrombus formation resulting from delayed neointimal coverage, spasms occurring at the distal end of the stent implantation site, positive remodeling of coronary arteries caused by local immune reaction to paclitaxel or rapamycin, and vascular endothelial damage induced by the polymer. For BMS, neointimal coverage begins within the first one month after stent implantation and almost completes in three months. For DES, sirolimus eluting stents (SES) for example, neointimal coverage is markedly delayed after stent implantation and the exposed stent struts may be largely attributable to the occurrence of late stent thrombosis.

On the other hand, everolimus eluting stents (EES), which have a thinner stent strut layer and improved polymer biocompatibility, it has been reported that earlier and more normal neointimal coverage can be achieved compared with other first-generation DESs, SES and paclitaxel eluting stents (PES). These findings suggest that coverage with vascular endothelium differs among different DES platforms. Optical coherence tomography (OCT) has a resolution of 15 to 20 μm, which is approximately 10 times higher than that of intravascular ultrasound (IVUS). It is therefore necessary to use OCT to accurately evaluate cross-sectional images of the stent struts covered with vascular endothelium. However, no studies have reported the results of continuous observation and evaluation of EES covered with endothelium.

Therefore, the investigators investigate time course of neointimal coverage of EES through detailed evaluation by OCT of neointimal coverage at 3, 6, and 12 months after stent implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 20 years old.
2. Indication of PCI.
3. To agree to review and record all the clinical course in this research protocol.
4. The patient who are eligible to receive dual antiplatelet therapy at least more than 6 month.
5. Informed concent with the document signed by the patients.

The patient have to correspond to all the above items at the time of registration.

Exclusion Criteria:

1. The patient who died during the research
2. The patient with Stent thrombosis during the research.
3. Previous history of pancytopenia, liver function, renal dysfunction, hypersensitive history of the drug.
4. Low ejection fraction (LVEF<=30%), an impaired liver function, and renal dysfunction (eGFR<=30)
5. The patient excluded from a safety of a thiazolidine derivative.

lesion exclusion criteria

1. left main artery
2. severe calcification
3. stent restenosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are percutaenous coronary intervention and stenting and eligible to receive dual antiplatelet therapy at least more than 6 month.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of neointimal coverage | 12 months
  The primary endpoint is to evaluate the neointimal coverage of XIENCE everolimus eluting stent (EES) in 12 month after stent implantation by Optical coherence tomography

SECONDARY OUTCOMES:
The percentage of neointimal coverage | 3 months
The percentage of neointimal coverage | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Toshiro Shinke, Principal Investigator — Kobe University Graduate School of Medicine
Locations (1):
- Kobe University Graduate School of Medicine, Kobe, Hyōgo, Japan